CLINICAL TRIAL: NCT01786018
Title: Allogeneic Transplantation After a Conditioning With Thiotepa, Busulfan and Fludarabin for the Treatment of Refractory/Early Relapsed Aggressive B-cell Non Hodgkin Lymphomas: a Phase II Multi-Center Trial
Brief Title: Thiotepa, Busulfan and Fludarabin for pt With Refractory/Early Relapsed Aggressive B-cell Non Hodgkin Lymphomas
Acronym: TBF
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera San Giovanni Battista (Other)
Responsible Party: Principal Investigator, Benedetto Bruno, MD, Azienda Ospedaliera San Giovanni Battista
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TBF2012
Record Dates: First submitted 2013-02-05; First posted 2013-02-07 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: B-cell Lymphoma Refractory
Keywords: Non Hodgkin lymphomas; Allogeneic Transplantation; Thiotepa; Busulfan; Fludarabin
MeSH Terms: interventions — Thiotepa; Busulfan; fludarabine phosphate; Transplantation; Hematocrit; Cytoreduction Surgical Procedures; Immunosuppression Therapy; Cyclosporine; Methotrexate; thymoglobulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): * Thiotepa 5 mg/kg/day on days -7, -6 (Total Dose 10 mg/kg)
  * Busulfan (i.v.) 3.2 mg/kg on days -5,-4,-3 (Total Dose 9.6 mg/kg)
  * Fludarabin: 50 mg/m2/day on days -5,-4,-3 (Total Dose 150 mg/m2)
  Interventions: Drug: Thiotepa; Drug: Busulfan; Drug: Fludarabin; Procedure: transplant (HCT); Radiation: Cytoreduction; Drug: Immunosuppression; Drug: Cyclosporine; Drug: Methotrexate; Drug: ATG; Procedure: Collection and infusions of Donor PBSC

INTERVENTIONS:
Drug: Thiotepa
  Other Names: TEPADINA®
Drug: Busulfan
  Other Names: BUSILVEX®
Drug: Fludarabin
  Other Names: FLUDARA®
Procedure: transplant (HCT) — Transplant will be PBSCs collected as per institutional standard. A portion of the PBSC product will be removed for DLI that is equivalent to 3x10^7 CD3 cells/kg recipient weight and cryopreserved.
Radiation: Cytoreduction — Cytoreduction and /or radiation therapy will be given by the referring physician or the attending physician as determined on clinical grounds or to meet eligibility requirements of the protocol for patients with advanced malignancy or to reduce tumor bulk. However, no intensive chemotherapy can be given within three weeks before conditioning.
Drug: Immunosuppression — Day -3. Commence cyclosporine at 5.0 mg/kg PO Q12 hours, continue to day +50 and then taper by 5% per week until day +180.
Drug: Cyclosporine — CSP is given based on adjusted body weight, at 5.0 mg/kg PO q12 hours from day -3.
  If there is nausea and vomiting at anytime during CSP treatment the drug should be given intravenously at the appropriate dose that was used to obtain a therapeutic level.
  See guidelines for PO to IV conversion below.
Drug: Methotrexate — Day 1 15 mg Days 3, 6, 11 10 mg m2 day IV for GVHD prevention
Drug: ATG — (FOR UNRELATED TRANSPLANTS ONLY) Days -3, -2: 2.5 mg /kg/day
  Other Names: Anti-Human Thymocyte Globulin
Procedure: Collection and infusions of Donor PBSC — Collection and infusions of Donor PBSC

SUMMARY:
The purpose of this study is to evaluate progression free survival, transplant-related morbidity (TRM) at day +100 and at +365, overall survival and incidence of acute and chronic GVHD in refractory/early relapsed aggressive B-cell non Hodgkin lymphomas patients treated with allogeneic Transplantation after a conditioning with Thiotepa, Busulfan and fludarabin.

DETAILED DESCRIPTION:
In the present study, it is hypothesised that patients with aggressive B cell lymphomas refractory to or relapsed early (within 12 months) after the completion of standard first-line immunoProtocol TBF2012 Version 1, 20 Nov 2012 9 chemotherapy can benefit from de-bulking salvage therapy (i.e. R-DHAP + bortezomib) followed by an allograft to improve progression-free survival.

Patient inclusion criteria

* Patients with refractory/relapsed aggressive B-cell non Hodgkin lymphomas after frontline therapy.
* Patients with stable disease or partial or complete remission (PET-negative) after salvage therapy
* Patients younger than 65 years old
* A fully HLA-identical sibling or matched unrelated donor is available. Patients with one antigen mismatched donors can be considered
* Patient must be competent to give consent

Patient exclusion criteria

* Patients treated with an autologous transplant as salvage therapy
* Patients with progressive lymphomas despite conventional therapies
* Patients with progressive lymphomas despite conventional therapies
* Uncontrolled CNS involvement with disease
* Fertile men or women unwilling to use contraceptive techniques during and for 12 months following treatment
* Females who are pregnant or breastfeeding
* Organ dysfunction defined as follows:

  * Cardiac function: ejection fraction <30% or uncontrolled cardiac failure
  * Pulmonary: DLCO <40% predicted
  * Liver function abnormalities: elevation of bilirubin to > 3 mg/dl and/or transaminases >4 the upper limit of normal
  * Renal: creatinine clearance <50 cc/min (24 hour urine Protocol TBF2012 Version 1, 20 Nov 2012 6 collection)
* Karnofsky performance score < 60%
* Patients with poorly controlled hypertension despite multiple antihypertensives
* Documented fungal disease that is progressive despite treatment
* Viral infections: HIV positive patients.
* Positive serology for Hepatitis B (HB) defined as a positive test for HBsAg. In addition, if negative for HBsAg but HBcAb positive (regardless of HBsAb status), a HBV DNA test will be performed and if positive the subject will be excluded.
* Positive serology for hepatitis C (HC) defined as a positive test for HCAb, in which case reflexively perform a HC RIBA immunoblot assay on the same sample to confirm the result
* Psychiatric disorders or psychosocial problems which in the opinion of the primary physician or Principal Investigator would place the patient at unacceptable risk from this regimen.
* Patients with active non-hematologic malignancies (except nonmelanoma skin cancers).
* Patients with a history of non-hematologic malignancies (except non-melanoma skin cancers) currently in a complete remission, who are less than 5 years from the time of complete remission, and have a >20% risk of disease recurrence. Donor inclusion criteria:
* Related or unrelated HLA identical donors who are in good health and have no contra-indication to donation. One antigen HLAmismatched (9/10 match) donors will also be considered.
* No contra-indication for the donor to collection by apheresis of mononuclear cells mobilized by G-CSF at a dose of 10-12 μg/kg of body weight.
* Donor must have adequate veins for leukapheresis or agree to placement of central venous catheter (femoral, subclavian). Donor exclusion criteria:
* Age < 18 years.
* Identical twin.
* Pregnancy.
* Infection with HIV.
* Inability to achieve adequate venous access.
* Known allergy to filgrastin (G-CSF).
* Current serious systemic illness.

Donor inclusion criteria:

* Related or unrelated HLA identical donors who are in good health and have no contra-indication to donation. One antigen HLAmismatched (9/10 match) donors will also be considered.
* No contra-indication for the donor to collection by apheresis of mononuclear cells mobilized by G-CSF at a dose of 10-12 μg/kg of body weight.
* Donor must have adequate veins for leukapheresis or agree to placement of central venous catheter (femoral, subclavian). Donor exclusion criteria:
* Age < 18 years.
* Identical twin.
* Pregnancy.
* Infection with HIV.
* Inability to achieve adequate venous access.
* Known allergy to filgrastin (G-CSF).
* Current serious systemic illness.

Donor inclusion criteria:

* Related or unrelated HLA identical donors who are in good health and have no contra-indication to donation. One antigen HLAmismatched (9/10 match) donors will also be considered.
* No contra-indication for the donor to collection by apheresis of mononuclear cells mobilized by G-CSF at a dose of 10-12 μg/kg of body weight.
* Donor must have adequate veins for leukapheresis or agree to placement of central venous catheter (femoral, subclavian). Donor exclusion criteria:
* Age < 18 years.
* Identical twin.
* Pregnancy.
* Infection with HIV.
* Inability to achieve adequate venous access.
* Known allergy to filgrastin (G-CSF).
* Current serious systemic illness.

ELIGIBILITY:
Patient inclusion criteria:

* Patients with refractory/relapsed aggressive B-cell non Hodgkin lymphomas after frontline therapy.
* Patients with stable disease or partial or complete remission (PET-negative) after salvage therapy
* Patients younger than 65 years old
* A fully HLA-identical sibling or matched unrelated donor is available. Patients with one antigen mismatched donors can be considered
* Patient must be competent to give consent.

Patient exclusion criteria:

* Patients treated with an autologous transplant as salvage therapy
* Patients with progressive lymphomas despite conventional therapies
* Patients with progressive lymphomas despite conventional therapies
* Uncontrolled CNS involvement with disease
* Fertile men or women unwilling to use contraceptive techniques during and for 12 months following treatment
* Females who are pregnant or breastfeeding
* Organ dysfunction defined as follows:

  * Cardiac function: ejection fraction <30% or uncontrolled cardiac failure
  * Pulmonary: DLCO <40% predicted
  * Liver function abnormalities: elevation of bilirubin to > 3 mg/dl and/or transaminases >4x the upper limit of normal
  * Renal: creatinine clearance <50 cc/min (24 hour urine collection)
* Karnofsky performance score < 60%
* Patients with poorly controlled hypertension despite multiple antihypertensives
* Documented fungal disease that is progressive despite treatment
* Viral infections: HIV positive patients.
* Positive serology for Hepatitis B (HB) defined as a positive test for HBsAg. In addition, if negative for HBsAg but HBcAb positive (regardless of HBsAb status), a HBV DNA test will be performed and if positive the subject will be excluded.
* Positive serology for hepatitis C (HC) defined as a positive test for HCAb, in which case reflexively perform a HC RIBA immunoblot assay on the same sample to confirm the result
* Psychiatric disorders or psychosocial problems which in the opinion of the primary physician or Principal Investigator would place the patient at unacceptable risk from this regimen.
* Patients with active non-hematologic malignancies (except non-melanoma skin cancers).
* Patients with a history of non-hematologic malignancies (except non-melanoma skin cancers) currently in a complete remission, who are less than 5 years from the time of complete remission, and have a >20% risk of disease recurrence.

Donor inclusion criteria:

* Related or unrelated HLA identical donors who are in good health and have no contra-indication to donation. One antigen HLA-mismatched (9/10 match) donors will also be considered.
* No contra-indication for the donor to collection by apheresis of mononuclear cells mobilized by G-CSF at a dose of 10-12 mg/kg of body weight.
* Donor must have adequate veins for leukapheresis or agree to placement of central venous catheter (femoral, subclavian).

Donor exclusion criteria:

* Age < 18 years.
* Identical twin.
* Pregnancy.
* Infection with HIV.
* Inability to achieve adequate venous access.
* Known allergy to filgrastin (G-CSF).
* Current serious systemic illness.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2013-02; Primary Completion 2015-02 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 2 years

SECONDARY OUTCOMES:
Transplant-related morbidity (TRM) at day +100 and at +365 | 1 year
Overall survival | 2 years
Incidence of acute and chronic GVHD | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Benedetto Bruno, MD, Principal Investigator — Divisione di Ematologia-Città della Salute e della Scienza di Torino
Locations (1):
- Città della Salute e della Scienza di Torino, Torino, Italy